CLINICAL TRIAL: NCT04257565
Title: Wheeling to Healing: Does Wheeled Knee Walker Use Improve Wound Healing, Improve Quality of Life and Decrease Risk of Contralateral Ulceration in People With Diabetic Foot Ulcers
Brief Title: Wheeling to Healing: A Novel Method for Improving Healing of Diabetic Foot Ulceration
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Collaborators: Saskatchewan Health Research Foundation (Other)
Responsible Party: Principal Investigator, Audrey Zucker-Levin, Professor, University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Bio1469
Record Dates: First submitted 2020-01-31; First posted 2020-02-06 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Diabetes Mellitus
Keywords: Foot Ulcer
MeSH Terms: conditions — Diabetes Mellitus; Foot Ulcer

STUDY DESIGN:
Intervention Model Description: randomized controlled clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): The Control Group will receive usual and customary care from their vascular specialist.
  Interventions: Other: Usual and Customary Care
- Intervention Group (Experimental): The Intervention Group will receive usual and customary care from their vascular specialist and they will be provided and trained to use the wheeled knee walker.
  Interventions: Device: Wheeled Knee Walker

INTERVENTIONS:
Device: Wheeled Knee Walker — The Wheeled Knee Walker allows total offloading of a healing limb and may diminish excessive force on the contralateral limb.
  Arms: Intervention Group
Other: Usual and Customary Care — This group will receive usual and customary care for treatment of their diabetic foot ulcer
  Arms: Control group

SUMMARY:
The increasing incidence of diabetes and high risk of amputation makes prevention and successful treatment of DFU of vital importance. A relatively new device, the wheeled knee walker, allows total offloading of the affected foot and, when compared to traditional walking aids such as crutches and walkers, requires significantly less physical exertion, is easier to use, and affords more stability. Its potential benefit to improve wound healing, impact physical function and quality of life in people with DFU is not yet known. Therefore, the goal of this research is to determine whether providing a wheeled knee walker to people with diabetic foot ulcers improves clinical outcomes and quality of life when compared to usual and customary care.

DETAILED DESCRIPTION:
The rate of diabetes in Saskatchewan is among the highest of all Canadian provinces with a prevalence of 8.5% in 2015 with an expected rise to 11.1% in 2025. Diabetic foot ulcers (DFU) are a common complication and the leading cause of lower limb amputation worldwide. Treatment for DFU include casts, braces, crutches and walkers to remove pressure (offload) from the ulcer. These interventions, when not rejected, foster a sedentary lifestyle which negatively impacts function and quality of life. Also, crutches and walkers may increase risk of ulceration of the sound foot as the arms are often not strong enough to support the body weight when stepping.

The wheeled knee walkers (WKW) is a relatively new walking aid that allows total offloading of one foot, requires less physical exertion, and is more stable than crutches or walkers. The purpose of this research is to determine if a WKW would improve wound healing, quality of life, and physical function while decreasing the risk of sound foot ulceration in people with DFU. To explore these objectives we will recruit people with DFU who are under the care of a vascular surgeon, perform standardized baseline measures for each objective, provide a WKW to half of the participants and then re-evaluate all objectives at 6 and 12 weeks. The results will help guide treatment and inform decision making to optimize care. Further, the project will establish an interdisciplinary collaborative research program for future projects to improve health and advance knowledge.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* currently under physician care for a DFU of one foot
* willing and able to sign informed consent
* cognitively functional
* have access to a telephone
* weigh no more than 300lbs as this is the weight limitation of the wheeled knee walker
* have at least one palpable foot pulse
* have a neuropathic plantar DFU corresponding to grade 1A (superficial, not extending to tendon, capsule, or bone) using the University of Texas Diabetic Foot Wound Classification System

Exclusion Criteria:

* coronary or cerebrovascular disease events within the past six months
* uncontrolled, severe medical conditions that place the subject at high risk for adverse events, including but not limited to severe congestive heart failure, angina pectoris, obstructive pulmonary disease
* uncontrolled neurologic or psychiatric disorders
* active infection
* significant ulcers or infections of both lower limbs
* those who have been wheelchair dependent prior to ulcer formation
* absence of pedal pulse
* any condition that would limit the ability to ambulate or stand without pain or discomfort, including but not limited to shortness of breath, fatigue, angina, severe arthritis
* medication use that causes impaired balance or judgment
* other circumstances at the investigators' and primary care providers' discretion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Wound Healing | 12 Weeks
  The wound will be measured using Image J, open source digital imaging software developed at the National Institutes of Health (NIH) to measure wound area of the target wound, in mm2 (the largest foot wound if multiple wounds are present). Image J software has been used specifically for the measurement of diabetic foot ulcers with very high inter- and intra-rater reliability (p=0.997 and 0.999 respectively) [1]. The wound will be traced on acetate paper using a fine permanent marker for use in Image J and a standard distance photograph of the wound will be taken to document wound bed characteristics after physician debridement to healthy granulating tissue or healthy bleeding tissue is reached [1, 2]. The physician will record depth at its greatest point using a probe at the time of debridement, assess wound condition (improving, stable, or deteriorating), and the presence or absence of undermining or tunneling. A completely healed wound has complete epithelialization.

SECONDARY OUTCOMES:
Quality of Life: The Diabetic Foot Ulcer Scale (DFS) | 12 weeks
  The Diabetic Foot Ulcer Scale (DFS) is a specific instrument designed to assess the impact of foot ulcers and their treatment on quality of life in people with Diabetes [3]. The DFS consists of 58 items grouped into 11 domains: leisure, physical health, daily activities, emotions, noncompliance, family, friends, positive attitude, treatment, satisfaction, and financial. The DFS has good internal consistency with adequate test-retest reliability and sensitivity to change in wound status over time indicating its appropriateness for use in clinical trials. DFS Items are scored by the individual using a five item (1-5) scale with higher scores indicating better quality of life. Score will be measured as an aggregate of all 58 items and individually in all 11 domains: Leisure, Physical health, Daily activities, Emotions, Noncompliance, Family, Friends, Treatment, Satisfaction, Positive Attitude, Financial.
Risk of ulceration of the sound foot | 12 weeks
  Risk of ulceration of the sound foot by measuring in-shoe foot force under the sound foot using a LoadSol® Insole (Novel Electronics Inc, St. Paul, MN) while the participant wears their 'usual' footwear. A 0.5 mm thick LoadSol® Insole corresponding to the participants shoe size will be placed between the sock and shoe of the sound foot prior to performing the 2-Minute Walk Test. The embedded grid of contact cells records the normal force between the plantar side of the foot and the shoe during activity. Foot force, in Newtons, will be measured during one minute of footfalls collected from 30 to 90 seconds of the 2-Minute Walk Test.
Physical Function | 12 weeks
  Physical function will be assessed by measuring distance walked (meters) in 2 minutes with Wheeled Knee Walker or Customary device. The 2-Minute Walk Test is a standardized and reliable clinically applicable method for quantifying physical function across and array of health conditions [4-6]. This test is safe in people with peripheral vascular diseases and heart disorders both of which can be precursors to DFU. It has also been proven to be reliable (intraclass coefficient = 0.94) for people with amputation due to diabetes [7]. Participants will be asked to walk in an unobstructed vacant hallway and to cover as much distance as safely possible in two minutes. The participant will wear their prescribed unloading protective footwear and use any prescribed assistive device for testing. They will be followed with a wheelchair in case rest is needed. The distance walked in two minutes will be measured and recorded using a distance measuring wheel.

CONTACTS AND LOCATIONS:
Overall Officials: Audrey R Zucker-Levin, PhD, Principal Investigator — University of Saskatchewan
Locations (1):
- University of Saskatchewan, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jeffcoate WJ, Musgrove AJ, Lincoln NB. Using image J to document healing in ulcers of the foot in diabetes. Int Wound J. 2017 Dec;14(6):1137-1139. doi: 10.1111/iwj.12769. Epub 2017 Jun 13. PMID 28612500
- [Background] Veves A, Murray HJ, Young MJ, Boulton AJ. The risk of foot ulceration in diabetic patients with high foot pressure: a prospective study. Diabetologia. 1992 Jul;35(7):660-3. doi: 10.1007/BF00400259. PMID 1644245
- [Background] Bohannon RW. Normative reference values for the two-minute walk test derived by meta-analysis. J Phys Ther Sci. 2017 Dec;29(12):2224-2227. doi: 10.1589/jpts.29.2224. Epub 2017 Dec 13. PMID 29643611
- [Background] Reid L, Thomson P, Besemann M, Dudek N. Going places: Does the two-minute walk test predict the six-minute walk test in lower extremity amputees? J Rehabil Med. 2015 Mar;47(3):256-61. doi: 10.2340/16501977-1916. PMID 25588644
- [Background] Brooks D, Hunter JP, Parsons J, Livsey E, Quirt J, Devlin M. Reliability of the two-minute walk test in individuals with transtibial amputation. Arch Phys Med Rehabil. 2002 Nov;83(11):1562-5. doi: 10.1053/apmr.2002.34600. PMID 12422326
- [Background] Lin SJ, Bose NH. Six-minute walk test in persons with transtibial amputation. Arch Phys Med Rehabil. 2008 Dec;89(12):2354-9. doi: 10.1016/j.apmr.2008.05.021. Epub 2008 Nov 1. PMID 18976979